CLINICAL TRIAL: NCT05451758
Title: Investigating the Role of Natural Environments in the Effectiveness of a Mindfulness-based Stress Reduction (MBSR) Programme
Brief Title: The Effectiveness of MBSR in Natural Environments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 150258786
Record Dates: First submitted 2022-06-24; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2017-04

CONDITIONS: Stress-related Problem
Keywords: Mindfulness; Stress
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Natural outdoor environment (Experimental): The park is a well-managed green space containing trees, shrubs, flower beds, lawns and a lake, and includes facilities such as benches, wooden bridges, a bandstand and monuments. The experiment was carried out in a location defined by planted areas containing shrubs and small trees, with some distant views.
  Interventions: Other: Mindfulness-based stress reduction (MBSR)
- Built outdoor environment (Experimental): A courtyard on the university campus was chosen as a built outdoor environment. The courtyard was surrounded by concrete and brick built settings, with no visible vegetation.
  Interventions: Other: Mindfulness-based stress reduction (MBSR)
- Indoor environment (Experimental): The indoor setting was a seminar room: a white painted room without windows in the basement of a university building. It contained chairs, a neutral coloured picture and no vegetation.
  Interventions: Other: Mindfulness-based stress reduction (MBSR)

INTERVENTIONS:
Other: Mindfulness-based stress reduction (MBSR) — The participants were asked to attend a brief version of the MBSR programme lasting six weeks. The intervention was a structured 6-week programme with groups of between 6 and 10 participants. Each weekly session lasted one hour and included mindfulness meditation/exercises and group discussion led by a qualified mindfulness instructor.

SUMMARY:
With the prescription of antidepressants at record levels, and a huge demand for psychological therapies, health and social care providers are interested in cost-effective interventions to improve wellbeing and to prevent mental health problems. At the same time, there is a renewed interest in complementary and alternative therapies, such as yoga, meditation practices, and aromatherapy to support psychological resilience and prevent mental illness.

Mindfulness practice has grown quickly as one such complementary and alternative approach to coping with certain forms of mental illness and symptoms of poor mental and physical health. The potential salutogenic benefits of mindfulness practice have been recognized, and mindfulness practice has received a great deal of attention as an intervention in a clinical/medical setting to address specific disorders (e.g. chronic pain or anxiety). The most widely used MBI is mindfulness-based stress reduction (MBSR), which offers an intensive 8-week programme (as well as shorter 4-6-week versions) involving a range of formal sitting and walking meditation, body scanning, mindful movement and informal mindfulness practices. Reviews of the effects and clinical effectiveness of MBSR indicate positive results in terms of the treatment of a range of different physiological and psychosocial conditions, including stress reduction and relief from emotional distress, depression and anxiety. Whilst this evidence demonstrates the significant mental health and wellbeing benefits of mindfulness-based interventions, there has been little research into combining mindfulness with restorative experiences, such as exposure to nature.

The aim of the study is to investigate whether the effectiveness of MBSR are enhanced when combined with a natural environment. The investigators hypothesise that MBSR in a natural environment results in greater nature connectedness than in a built outdoor or an indoor environment (hypothesis 1). It is also hypothesised that MBSR achieves the best mental health and wellbeing outcomes when conducted in a natural environment (hypothesis 2).

DETAILED DESCRIPTION:
The experimental design combined MBSR with an environmental condition. Participants were randomly assigned to brief MBSR in one of the three different environments (i.e., natural outdoor environment, built outdoor environment and indoor environment). All participants were asked to attend the brief MBSR programme for 6 weeks with 1-hour sessions. The weekly MBSR session included sitting and body scanning meditation, mindfulness exercises and group discussion led by a qualified mindfulness facilitator. During the experiment, participants were asked to complete the same questions in DASS-21 four times: baseline, after 3 weeks, after 6 weeks (at the completion of the 6-week MBSR) and one-month follow-up. In addition, participants who attended at least five of the six MBSR sessions were invited to donate their hair samples to measure the change of their stress level.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Students and staff at the University of Sheffield

Exclusion Criteria:

* Having severe and enduring mental health conditions (i.e. people currently receiving treatment for such conditions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Change in positive and negative emotions | Change in PANAS from baseline to one month after the completion of the 6-week MBSR
  The Positive and Negative Affect Schedule (PANAS) measures hedonic wellbeing, eliciting respondent's current state across a wide variety of emotions. The PANAS contains two 10-item subscales designed to measure positive feelings (i.e. interested, excited, strong, enthusiastic, proud, alert, inspired, attentive, determined and active), and negative feelings (i.e. distressed, upset, guilty, scared, hostile, irritated, ashamed, nervous, jittery and afraid). Respondents were asked how much they felt each of the 20 emotions (1= not at all, 5= extremely). Scores ranged from 10 to 50 with higher scores indicating higher levels of positive or negative feelings
Change in depression, anxiety and stress | Change in DASS-21 from baseline to one month after the completion of the 6-week MBSR
  Depression Anxiety Stress Scales (DASS-21) contains 21 psychological questions related to the symptoms of depression, anxiety and stress (Lovibond and Lovibond, 1995; Antony et al., 1998). The DASS-21 contains three self-report subscales with seven phrases that describe how respondents felt in the past week on a four-point scale (0= never, 3= almost always): e.g. Depression ("I felt that I had nothing to look forward to"); e.g. Anxiety ("I was worried about situations in which I might panic and make a fool of myself"); and e.g. Stress ("I found it difficult to relax"). Scores ranged from 0 to 42 with higher scores indicating higher levels of depression, anxiety and stress.
Change in hair cortisol concentration (HCC) | Change in HCC from baseline to one month after the completion of the 6-week MBSR
  Hair cortisol concentration (HCC) is used as a marker of chronic stress. Cortisol is commonly known as the stress hormone because it is released via the hypothalamic-pituitary-adrenal (HPA) in higher doses under stressful conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Yeong Choe, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Department of Landscape Architecture, University of Sheffield, Sheffield, United Kingdom